CLINICAL TRIAL: NCT05620303
Title: A Healthy Lifestyle-based Randomized Controlled Trial on 24-h Movement Behaviors and Adherence to the Mediterranean Diet in Schoolchildren - The Archena Infancia Saludable Project: A Protocol Study
Brief Title: 24-h Movement Behaviors and Adherence to the Mediterranean Diet in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Castilla-La Mancha (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: UCLMCFE00085
Record Dates: First submitted 2022-11-09; First posted 2022-11-17 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Mediterranean Diet; Physical Activity; Sedentary Time; Sleep
Keywords: Physical activity; Sedentary behavior; Screen time; Sleep duration; Movement guidelines
MeSH Terms: conditions — Motor Activity; Sedentary Behavior | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Cluster randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Experimental)
  Interventions: Other: Exercise
- Control group (No Intervention)

INTERVENTIONS:
Other: Exercise — Parents/guardians will receive three different contents weekly (i.e., infographics, video recipes, information pills, or videos) each week related to 24-h movement behaviors (i.e., PA, sedentary behavior, sleep duration) or Mediterranean Diet for 36 weeks.
  Arms: Exercise group

SUMMARY:
The purpose of this study is to determine the effects of the Archena Infancia Saludable project on adherence to MD and 24-h movement behaviors in schoolchildren

ELIGIBILITY:
Inclusion Criteria:

Schoolchildren aged 6-13 years will be eligible

Exclusion Criteria:

* Participants with any pathology that contraindicate exercise or that request special attention.
* Participants under pharmacological treatment that prevent them from receiving the contents of the activities of the program.
* Participants or parents/legal guardians presenting Spanish learning difficulties.
* Participants do not authorized by the parents/guardians to be included in the research project.
* Participants do not agree to take part in the research project.

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 154 (Actual)
Dates: Start 2022-12-02 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Adherence to the Mediterranean diet | From baseline to 36 weeks later
  To assess the adherence to the Mediterranean Diet, the Mediterranean Diet Quality Index for Children and Teenagers (KIDMED) index will be used.
24-h movement behaviors (accelerometers) sedentary time | From baseline to 36 weeks later
  A tri-axial accelerometer (Actigraph GT3x, Pensacola, FL, USA) will be used to assess sedentary time over seven consecutive days.
24-h movement behaviors (self-reported) | From baseline to 36 weeks later
  Self-report of physical activity levels and sedentary behaviors in youth will assessed by the Youth Activity Profile - Spain. In this questionnaire, a rating scale is used with a score from 1 to 5 in which, in the first two sections, "1" indicates low intensity and frequency of physical activity and "5" indicates high intensity and frequency of physical activity; while, in the third section, "1" indicates a low amount of sedentary behaviors and "5" an excess of them.
24-h movement behaviors (accelerometers) physical activity | From baseline to 36 weeks later
  A tri-axial accelerometer (Actigraph GT3x, Pensacola, FL, USA) will be used to assess physical activity over seven consecutive days.
24-h movement behaviors (accelerometers) sleep duration | From baseline to 36 weeks later.
  A tri-axial accelerometer (Actigraph GT3x, Pensacola, FL, USA) will be used to assess sleep duration over seven consecutive days.

SECONDARY OUTCOMES:
Anthropometrics measurements | From baseline to 36 weeks later
  The body weight of the schoolchildren will be measured using an electronic scale (with an accuracy of 0.1 kg) (Tanita BC-545, Tokyo, Japan), while height will be determined by a portable height rod with an accuracy of 0.1 cm (Leicester Tanita HR 001, Tokyo, Japan). Body mass index (BMI) will be calculated by dividing body weight (in kg) by the height (in squared meters). Furthermore, BMI z-score will be computed by the WHO age-specific and sex-specific thresholds.
Active transportation | From baseline to 36 weeks later
  Active transportation to and from school is evaluated by a self-reported questionnaire (Mode and Frequency of Commuting To and From School Questionnaire). Participants were categorized as "active" if reported: ≥2 active travel days out of 5 school days (questions #1 and #2) and ≥ 4 active travel trips out of 10 school trips per week (question #3). The usual mode of commuting to/from school was categorized as active when participants reported ≥ 1 active travel per day out of 2 daily school trips (question #4). Those who were not categorized as "active commuting" were categorized as "passive commuting" users.
Resting blood pressure | From baseline to 36 weeks later
  Resting blood pressure will be measured using an automated blood pressure monitor with a fittingly sized cuff (Omrom® EVOLV HEM-7600T-E, Health-care Co, Kyoto, Japan). First, schoolchildren will be seated in a quiet room for 10 min with their feet on the ground and their back supported. Two readings will be taken, with the second blood pressure reading taken five min after the first. The average of the two measurements for systolic blood pressure and diastolic blood pressure will be retained. Subsequently, mean arterial pressure will be computed by the following formula: diastolic blood pressure + [0.333 × (systolic blood pressure - diastolic blood pressure)].
Sleep disorders | From baseline to 36 weeks later
  Sleep disorders will be evaluated by the BEARS (B = Bedtime Issues, E = Excessive Daytime Sleepiness, A = Night Awakenings, R = Regularity and Duration of Sleep, S = Snoring) scale. Any questions that are answered positively indicate a sleep problem.
Health-related quality of life | From baseline to 36 weeks later
  Health-related quality of life will be measured by Child Health Utility 9D (CHU9D). The CHU9D consists of 9 dimensions: worried, sad, pain, tired, annoyed, schoolwork/homework, sleep, daily routine, ability to join in activities with five different levels representing increasing levels of severity within each dimension. Furthermore, CHU9D scores will be used in cost-utility analyses.
Self-reported physical fitness | From baseline to 36 weeks later
  Self-reported physical fitness will be assessed by the International Fitness Scale (IFIS), which is composed of a 5-point Likert-scale items asking about the children' perceived global physical fitness, cardiorespiratory fitness, muscular fitness, speed-agility, and flexibility in comparison with their counterparts' physical fitness (very poor (1), poor (2), average (3), good (4), and very good (5)).
Parents'/guardians' perception of their children's body mass index status | From baseline to 36 weeks later
  This outcome will be evaluated with the following question: "In relation to his/her height, which of the following options best describes your child's weight: 1) substantially above normal, 2) slightly above normal, 3) normal, 4) below normal?".
Academic performance | From baseline to 36 weeks later.
  Academic records will be provided at the end of the academic year by the school. Firstly, academic performance will be evaluated according to the grade obtained in Language, Mathematics, Language and Mathematics (combined), English, as well as the grade point average of these three subjects. Secondly, academic performance will be assessed by computing the grade point average of all the subjects taken by the children.

OTHER OUTCOMES:
24-h movement behaviors (self-reported) parents/guardians | From baseline to 36 weeks later.
  The level of physical activity and sitting time will be assessed by the International Physical Activity Questionnaire-short form (IPAQ-SF).
Adherence to the Mediterranean diet (parents/guardians) | From baseline to 36 weeks later.
  Parents/guardians will be also administered a 17-item Mediterranean dietary questionnaire, a modified version of the previously validated questionnaire used in the PREDIMED trial designed to assess adherence to Mediterranean Diet. Meeting with each of the 17 items relating to characteristic food habits will be scored with zero or one point. Therefore, the total score will range from 0 to 17 points, with 0 points denoting no adherence to the MD and 17 meaning maximum adherence to the Mediterranean Diet.
Anthropometrics measurements (parents/guardians) | From baseline to 36 weeks later.
  The body weight and body height of the parents/guardians will be self-reported. Body mass index (BMI) will be computed by dividing body weight (in kg) by the height (in squared meters).

CONTACTS AND LOCATIONS:
Locations (1):
- Colegio El Ope, Murcia, Spain